CLINICAL TRIAL: NCT03775746
Title: Can Very Low Dose Rivaroxaban in Addition to Dual Antiplatelet Therapy (DAPT) Improve Thrombotic Status in Acute Coronray Syndrome (ACS) ACS
Acronym: VaLiDate-R
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD2018-41
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Rivaroxaban; Tablets; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clopidogrel with Rivaroxaban (Experimental): Clopidogrel 75mg o.d. and Rivaroxaban 2.5mg b.i.d.
  Interventions: Drug: Clopidogrel 75Mg Tablet; Drug: Rivaroxaban 2.5Mg Tablet
- Clopidogrel (Active Comparator): Clopidogrel 75mg o.d.
  Interventions: Drug: Clopidogrel 75Mg Tablet
- Ticagrelor (Active Comparator): Ticagrelor 90mg b.i.d.
  Interventions: Drug: Ticagrelor 90Mg Tablet

INTERVENTIONS:
Drug: Clopidogrel 75Mg Tablet — Prevention of atherothrombotic events in percutaneous coronary intervention (adjunct with aspirin) in patients not already on clopidogrel
  Other Names: EU/1/08/465/001
  Arms: Clopidogrel; Clopidogrel with Rivaroxaban
Drug: Rivaroxaban 2.5Mg Tablet — Prophylaxis of atherothrombotic events following an acute coronary syndrome with elevated cardiac biomarkers (in combination with aspirin alone or aspirin and clopidogrel)
  Other Names: EU/1/08/472/025-035; EU/1/08/472/041; EU/1/08/472/046-047
  Arms: Clopidogrel with Rivaroxaban
Drug: Ticagrelor 90Mg Tablet — Prevention of atherothrombotic events in patients with acute coronary syndrome [in combination with aspirin]
  Other Names: EU/1/10/655/007-011
  Arms: Ticagrelor

SUMMARY:
A prospective, randomised, open label study of 3 clinically licensed treatments for ACS to assess the effects of these treatments on blood tests of endogenous fibrinolysis. 50 patients will be randomised to each of the 3 treatment arms in 1:1:1 ratio. Patients will receive the randomised treatment for 1 month after their index admission with ACS.

DETAILED DESCRIPTION:
Heart attacks are caused by a blood clot occurring in a blood vessel (artery) which supplies blood to the heart. Such a clot can build up and block the blood flow, depriving part of the heart muscle of oxygen and blood, causing transient or permanent damage to the heart muscle.

The standard treatment for a heart attack is two blood thinning medications combined, every day, to reduce the risk of further blood clots forming and to prevent another heart attack. The highest risk of another heart attack is in the next 30 days after the first heart attack.

However, despite two blood thinners combined, some patients still go on to have another clot (heart attack or stroke or death) and this can be life threatening. Earlier research has shown that through a blood test, it is possible to identify patients who remain at increased risk of further clots and who may benefit from further blood thinners to reduce the risk of further heart attack, stroke and death in the next 30 days.

The aim of this study is to test which of 3 blood thinning treatment options (all already in widespread clinical use) is best for patients to reduce further blood clots, in particular the addition of low dose rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years or over
2. Have a diagnosis of acute coronary syndrome requiring treatment with dual antiplatelet therapy
3. Be willing and able to understand the Participant Information Sheet and provide informed consent
4. Agree to comply with the drawing of blood samples for the assessments
5. Not meet any of the exclusion criteria below

Exclusion Criteria:

1. Male and female participants aged < 18 years of age.
2. Patient unwilling or unable to give informed consent
3. Patients who might be pregnant or are breast-feeding
4. Active clinically significant bleeding
5. Patient who, in the opinion of the investigator, has condition considered to be a significant risk for major bleeding (such as current or recent gastrointestinal ulceration, presence of malignant neoplasm at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial haemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities)
6. Hepatic disease associated with coagulopathy and clinically relevant bleeding risk including cirrhotic patients with Child Pugh B and C
7. Patient with any contraindications to use of antiplatelet agents or anticoagulants
8. Hypersensitivity to the active substance or to any of the excipients listed in section 6.1 of Summary of Product Characteristics (SmPC) of Rivaroxaban
9. Concomitant treatment with any other anticoagulants e.g. unfractionated heparin (UFH), low molecular weight heparins (enoxaparin, dalteparin, etc.), heparin derivatives (fondaparinux, etc.), oral anticoagulants (warfarin, dabigatran etexilate, apixaban etc.) except under specific circumstances of switching anticoagulant therapy or when UFH is given at doses necessary to maintain an open central venous or arterial catheter
10. Concomitant treatment of ACS with antiplatelet therapy in patients with a prior stroke or a transient ischaemic attack (TIA)
11. Patient with ongoing active alcohol or substance abuse or demonstrates signs or clinical features of active substance abuse.
12. Patient with any major bleeding diathesis or blood dyscrasia at baseline (platelets<70 x 109/l, Hb<80 g/l, INR>1.4, APTT> x 2UNL, leucocyte count< 3.5x 109/l, neutrophil count<1x 109/l)
13. Patient currently enrolled in an investigational drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The change in Lysis Time (LT) in the three treatment groups assessed using the GTT from admission to follow-up at 30 days | 30 days
  To investigate, in patients with recent acute coronary syndrome and who have impaired endogenous fibrinolysis, whether the addition of low dose rivaroxaban to DAPT can improve endogenous thrombotic and fibrinolytic status

SECONDARY OUTCOMES:
Frequency of further angioplasty | 6 months
  Clinical events including re-intervention
Frequency of further heart attack, stroke or death | 6 months
  Incidence of further major adverse cardiac events

CONTACTS AND LOCATIONS:
Locations (1):
- East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gue YX, Kanji R, Wellsted DM, Srinivasan M, Wyatt S, Gorog DA. Rationale and design of "Can Very Low Dose Rivaroxaban (VLDR) in addition to dual antiplatelet therapy improve thrombotic status in acute coronary syndrome (VaLiDate-R)" study : A randomised trial modulating endogenous fibrinolysis in patients with acute coronary syndrome. J Thromb Thrombolysis. 2020 Feb;49(2):192-198. doi: 10.1007/s11239-019-02014-5. PMID 31872349